CLINICAL TRIAL: NCT01279239
Title: Establishing 1H Nuclear Magnetic Resonance (NMR) Based Metabonomics Fingerprinting Profile for Severe Poly Trauma Patients
Brief Title: Metabonomics Fingerprinting of Multiple Trauma
Status: Completed | Type: Observational
Sponsor: Sichuan Academy of Medical Sciences (Other)
Responsible Party: Hua Jiang/Deputy Chief Surgeon, Sichuan Academy of Medical Sciences, Sichuan Provincial People's Hospital
Other Study IDs: META-LAB-10-07-003C-02
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Trauma
Keywords: Poly Trauma; Metabonomics; NMR; MOF
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma from peripheral blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Poly trauma: 20 Patients suffering from poly trauma who meet inclusion criteria would be recruited
- Healthy control: 20 healthy volunteers would be recruited to obtain basal metabonomics fingerprinting

SUMMARY:
The aim of this study is to establish plasma metabonomics fingerprinting atlas for severe multiple trauma patient using 1H nuclear magnetic resonance (NMR) based metabonomics methodology and advanced mathematics tools.

DETAILED DESCRIPTION:
Metabonomics is a set of measurements of the dynamic metabolic responses of living systems to stimuli or modifications. This field of study developed from the application of nuclear magnetic resonance (NMR) spectroscopy and mass spectrometry as tools for the study of complex biofluids. Metabonomics is one of the emerging fields of systemic biology researches concerned with the high-throughput identification, quantification and characterization of small molecule metabolites. A metabonomics fingerprinting can be defined as the complete complement of all small molecule (<1500 Da) metabolites found in a specific cell, body fluid, organ or organism.

Severe poly trauma involves complex injuries that consist of multiple pathological mechanisms involving cytotoxic, oxidation stress and immune-endocrine. The complexity of the pathological physiology and biochemistry process are determined not only by the initial mechanical assault, but also by secondary processes including abnormality of inflammation regulation, ischemia, anoxia, free-radical formation, and immune dysfunction that occur over hours and days following the injury. For the clinical perspective, one of the key difficulties is to identify the most at-risk patients who could develop multiple organ failures and consequently death.

This study aims to establish the dynamics of NMR-based metabonomics fingerprinting of severe multi-trauma patients in order to provide a possible multiple organs failure (MOF) or death event prediction.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-50 years
* Poly trauma
* Injury Severity Score (ISS)>16 and Acute Physiology And Chronic Health Evaluation(APACHE)II>10

Exclusion Criteria:

* With comorbidity (Diabetes,Hyperthyroidism or primary organ dysfunction )
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are suffering from poly trauma.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mortality at hospitalization | Death events from admission to discharge(up to 10 weeks)

SECONDARY OUTCOMES:
Multi Organ Failure(MOF) | MOF events occurence from admission to discharge(up to 10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, M.D, Study Chair — Sichuan Academy of Medical Sciences; Zhi-Yuan Zhou, M.S, Principal Investigator — Sichuan Academy of Medical Sciences; Ming-Wei Sun, M.D, Principal Investigator — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan Academy of Medical Sciences, Sichuan Provincial Hospital, Dept. Trauma Surgery, Chengdu, Sichuan, China